CLINICAL TRIAL: NCT01850589
Title: Comparison of Conservative and Aggressive Smoking Cessation Treatment Strategies in a Vascular Surgery Office Practice
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Use of bupropion with counseling works better to help patients quit smoking.
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Jonathan Deitch, Program Director, Vascular Surgery, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11-001
Record Dates: First submitted 2013-04-08; First posted 2013-05-09 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — halofantrine; Bupropion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative Therapy (Other): Conservative therapy:
  Subjects counseled by vascular attending/fellow during office appointment to stop smoking.
  Counseling consists of:
  Self-help materials including "Smart Move: A Stop Smoking Guide" from the American Cancer Society A brief educational discussion on the benefits of smoking cessation.
  Patients randomized to Group 1 will be offered adjunctive treatment with nicotine replacement therapy at no cost.
  Interventions: Other: Aggressive Therapy
- Aggressive Therapy (Other): 8 week comprehensive smoking cessation and pharmacotherapy program consisting of:
  * One hour group counseling sessions, focusing on patient education and behavior modification.
  * Behavior modifications including recognition; coping skills; stress management; and relapse prevention skills.
  * Counseling including information on nutrition, exercise, and chemical dependency.
  Counseling sessions will be held 256C Mason Avenue. Pharmacotherapy adjuncts offered at no cost are as follows: Chantix (varenicline) GlaxoSmithKline, Zyban (bupropion) Pfizer,and Nicoderm/Nicorette (nicotine nasal spray, inhaler, transdermal patches and gum) GlaxoSmithKline.
  Interventions: Other: Aggressive Therapy

INTERVENTIONS:
Other: Aggressive Therapy — Pharmacotherapy adjuncts offered at no cost are as follows:
  * Chantix (varenicline) GlaxoSmithKline,
  * Zyban (bupropion) Pfizer,and Nicoderm/Nicorette (nicotine nasal spray, inhaler, transdermal patches and gum) GlaxoSmithKline.
  Other Names: GlaxoSmithKline, Zyban,Nicoderm/Nicroette GlaxoSmithKline.

SUMMARY:
The aim of this study is to prove that the use of Bupropion with counseling works better than counseling alone for patients to quit smoking. The belief is that overall, there is a small percentage of patients who quit smoking all together.

DETAILED DESCRIPTION:
The objective of the current investigation is to evaluate the effectiveness of an intensive verses conservative smoking cessation program in patients with peripheral arterial disease in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with confirmed peripheral arterial disease (PAD), defined as at least one of the following criteria, during the initial Vascular Surgery Office exam and review of the patient's medical record:

   1. Ankle-brachial index of <.90 in at least 1 lower extremity.
   2. Toe-brachial index of <.60
   3. Objective evidence of arterial occlusive disease in 1 lower extremity by duplex ultrasonography, magnetic resonance angiography or computed tomographic angiography
   4. prior leg arterial revascularization or amputation due to PAD
2. Patients have to smoke with a minimum of 10 cigarettes per day for a minimum of 5 years.
3. Patients must be able to give informed written consent and be at least 18 years of age.

Exclusion Criteria:

1. Pregnant women: Smoking Cessation Program medication Chantix (varenicline), Zyban (bupropion) has been shown to cause decreased fertility and decrease fetal weight in animal study offspring.
2. Patients less than 18 years of age: Safe and effective use in children has not been established with Chantix (varenicline) and Zyban (bupropion). These medications are not approved for use in individuals less than 18 years of old.
3. Patients with a history of a seizure disorder. Zyban (bupropion) is contraindicated in patients with preexisting seizure disorder.
4. Patients with a history of anorexia nervosa or bulimia nervosa. Patients with these eating disorders have been shown to have an increased incidence of seizures and Zyban (bupropion) is contraindicated in patients with a history or anorexia nervosa and bulimia nervosa.
5. The use bupropion concomitantly with monoamine oxidase inhibitors (MAOIs), including drugs with MAOI-like activity is contraindicated. Studies with animals indicate that bupropion-induced adverse reaction and toxicity appear to be enhanced by these medications.
6. Patients with renal insufficiency;defined as having a Creatinine Clearance (CrCl) <=50mL/min. Chantix is substantially excreted by the kidneys and the risk of toxic reactions are greater in patients with impaired renal function. Creatinine Clearance =[(140-age(yr)]*weight(kg)]/[72*serumCr(mg/dL)].
7. Patients with hepatic insufficiency; defined as having elevated liver function tests (serum aminotransferases) greater than 1.5 baseline. Zyban is metabolized in the liver. Half-lives of bupropion and/or its major metabolites are prolonged in patients with liver disease.
8. Patients with vascular pathology other than PAD (Carotid atherosclerosis, abdominal aortic aneurysms, venous insufficiency).
9. Subjects with a history of psychiatric illness requiring current treatment with psychoactive medications, a history of dependence on alcohol or non nicotine substance in the past year or current use of tobacco products other than cigarettes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Deitch, MD, Principal Investigator — North Shore- LIJ Health System (SIUH)
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Conserative Therapy: Patients will be counseled by the vascular attending/fellow during their office appointment to stop smoking. Counseling will consist of a self-help materials including "Smart Move: A Stop Smoking Guide" from the American Cancer Society and a brief educational discussion on the benefits of smoking cessation. Patients randomized to Group 1 will be offered adjunctive treatment with nicotine replacement therapy at no cost.
- Aggressive Therapy: 8 week comprehensive smoking cessation and pharmacotherapy program consisting of:
  * 8 one hour group counseling sessions focusing on patient education and behavior modification.
  * Behavior modifications include cue recognition; coping skills; stress management; and relapse prevention skills.
  * Counseling includes information on nutrition, exercise, and chemical dependency.
  All counseling sessions will be held at 256C Mason Avenue. Pharmacotherapy adjuncts offered at no cost are as follows:
  * Chantix (varenicline) GlaxoSmithKline,
  * Zyban (bupropion) Pfizer
  * Nicoderm/Nicorette (nicotine nasal spray, inhaler, transdermal patches and gum) GlaxoSmithKline.
Period: Overall Study
Arm/Group | Conserative Therapy | Aggressive Therapy
Started | 22 | 22
Completed | 14 | 22
Not Completed | 8 | 0
Not completed — Withdrawal by Subject | 8 | 0

BASELINE CHARACTERISTICS:
Population: There were a total of 44 subjects enrolled. 36 successfully completed the therapy. 14 subjects: Conservative management, 22 subjects: Aggressive Managment. 8 subjects withdrew from the study.
Groups:
- Conserative Therapy: Patients counseled by the vascular attending/fellow during office appointment to stop smoking. Counseling consists of self-help materials including "Smart Move: A Stop Smoking Guide" from the American Cancer Society and a brief educational discussion on the benefits of smoking cessation. Patients randomized to Group 1 will be offered adjunctive treatment with nicotine replacement therapy at no cost.
- Aggressive Therapy: 8 week comprehensive smoking cessation and pharmacotherapy program consisting of:
  * One hour group counseling sessions, focusing on patient education and behavior modification.
  * Behavior modifications including recognition; coping skills; stress management; and relapse prevention skills.
  * Counseling including information on nutrition, exercise, and chemical dependency.
  Counseling sessions will be held 256C Mason Avenue. Pharmacotherapy adjuncts offered at no cost are as follows: Chantix (varenicline) GlaxoSmithKline, Zyban (bupropion) Pfizer,and Nicoderm/Nicorette (nicotine nasal spray, inhaler, transdermal patches and gum) GlaxoSmithKline.
  Varenicline, Bupropion,and nicotine nasal spray, inhaler, transdermal patches and gum: Pharmacotherapy adjuncts offered at no cost are as follows:
  * Chantix (varenicline) GlaxoSmithKline,
  * Zyban (bupropion) Pfizer,and Nicoderm/Nicorette (nicotine nasal spray, inhaler, transdermal patches and gum) GlaxoSmithKline.
- Total: Total of all reporting groups
Arm/Group | Conserative Therapy | Aggressive Therapy | Total
Number analyzed (Participants) | 14 | 22 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 22 | 36
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: Participants] — Gender data was not collected in this study.
  Participants
    Unspecified Gender | 14 | 22 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Smoking Cessation at 12 Months
Description: Conservative vs. aggressive smoking strategies in treating smoking cessation.
Time Frame: 12 months
Population: Mean follow up was 7.3 months
Measure: Number; unit: Participants
Arm/Group | Conserative Therapy | Aggressive Therapy
Number analyzed (Participants) | 14 | 22
Participants | 4 | 10

ADVERSE EVENTS:
Arm/Group | Conserative Therapy | Aggressive Therapy
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No